CLINICAL TRIAL: NCT06040125
Title: Debunking the Frailty-sarcopenIa-ADT Axis in mEtastatic Prostate canceR With multiComponent Exercise: The FIERCE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-109
Record Dates: First submitted 2023-08-10; First posted 2023-09-15 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: PROSTATE CANCER; Metastatic Prostate Cancer; Metastatic Prostate Carcinoma
Keywords: Prostate Cancer; Metastatic Prostate Cancer; Metastatic Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants will partake in a 16-week supervised exercise program.
  Interventions: Behavioral: Supervised Circuit Training
- Attention Control Group (Experimental): Participants will continue with their normal daily activities.
  Interventions: Behavioral: Supervised Circuit Training

INTERVENTIONS:
Behavioral: Supervised Circuit Training — 16-week, multicomponent exercise intervention comprised of sessions supervised by certified exercise oncology trainer and home-based, self-directed aerobic exercises. Stationary bike and accelerometer (activity/heart rate monitor) will be provided.

SUMMARY:
The purpose of this study is to determine whether a 16-week supervised, clinic-based circuit training intervention utilizing resistance and functional exercises and self-directed aerobic exercise will improve frailty and sarcopenic status and disease progression outcomes among pre-frail/frail metastatic prostate cancer patients receiving androgen deprivation therapy (ADT).

The names of the study intervention involved in this study is:

• Supervised circuit training (aerobic and resistance exercise regimen)

DETAILED DESCRIPTION:
This research study is a pilot, randomized control study, which is the first-time investigators are examining this intervention in this setting.

Participants will be randomized into one of two study groups: Exercise Group versus Attention Control Group. Randomization means a participant is placed into a group by chance.

The research study procedures include screening for eligibility, study treatment, including extensive evaluations of fitness, physical health and strength, blood tests, muscle biopsy, surveys, and follow-up visits.

Participation in this research study is expected to last about 16 weeks.

It is expected that about 80 people will take part in this research study.

The Prostate Cancer Foundation is providing funding for this research study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign informed consent prior to any study-related procedures.
* Diagnosed with metastatic prostate cancer.
* Aged ≥18 years; due to the rarity of the disease in those <18 years, this age bracket will not be included.
* Have been receiving androgen deprivation (either with or without androgen receptor targeted treatment) for at least one month and expect to remain on their treatment for at least 4 months.
* Are pre-frail or frail as indicated by the FRAIL scale (a score of 1-2 = pre-frail; 3-5 = frail).
* Have physician's clearance to participate in exercise.
* Speak English.
* Participate in less than 2 structured resistance exercise sessions per week over the last 4 months.
* Participate in less than or equal to 60 minutes of moderate-to-vigorous aerobic exercise per week over the last month.
* Willing to travel to Dana-Farber Cancer Institute for necessary data collection and exercise sessions.

Exclusion Criteria:

* Receiving chemotherapy. This study is exclusively targeting androgen deprivation therapy-related effects.
* Have unstable bone lesions. In general patients with severely symptomatic/unstable bone lesions due to bone metastases are at a higher risk of fractures.
* Complete 2 or more structured resistance exercise sessions per week over the last 4 months and participate in more than 60 minutes of moderate-to-vigorous aerobic exercise per week over the last month. Excess additional exercise is a confounding factor in assessing the effect of the current exercise program.
* Unstable comorbidities that prevent participation in moderate-to-vigorous intensity exercise. Patients with unstable comorbidities likely require supervised exercise for safety, and part of this study involves unsupervised exercise; therefore, for safety reasons, these persons are excluded.
* Patients receiving treatment for other active malignancies (except basal cell carcinoma). This study is exclusively targeting androgen deprivation therapy-related effects.
* Subjects who in the opinion of the investigators may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Circulating Inflammation for Exercise Group | Baseline (week 0) and Post-intervention (week 17)
  Assessed by change in systemic inflammatory biomarkers through blood analysis (ul/ml).
Frailty | Baseline (week 0) and Post-intervention (week 17)
  This will be assessed by the Fried Frailty Phenotype, which measures participant ratings on a five-characteristic scale and will be totaled for an overall frailty score of 1-2, identified as prefail, or ≥3, identified as frail. Participants will receive a score of 1 (experience characteristic) or 0 (do not experience) for each characteristic.

SECONDARY OUTCOMES:
Sarcopenia | Baseline (week 0) and Post-intervention (week 17)
  A sarcopenia score of ≤10.75 kg/m2, as assessed by computed tomography (CT), will be the cut point used for identifying muscle loss = 1 point.
Skeletal Muscle Biomarkers - myokines | Baseline (week 0) and Post-intervention (week 17)
  Assessed from muscle biopsy specimens of the vastus lateralis (ul/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Wilson RL, Vulczak A, Morgans AK, Norris M, Greer J, Votta J, Vamvini M, Einstein DJ, Uno H, Rosenthal M, Vander Heiden MG, Dieli-Conwright CM. Design of debunking the frailty-sarcopenia-ADT axis in metastatic prostate cancer with multicomponent exercise: the FIERCE trial protocol. Front Sports Act Living. 2025 Oct 23;7:1602123. doi: 10.3389/fspor.2025.1602123. eCollection 2025. PMID 41210271